CLINICAL TRIAL: NCT03752216
Title: Longitudinal Study Evaluating in Real Life the Tolerability of Niraparib in Maintenance After Platine-based Chemotherapy for Patients with Ovarian Cancer Late Relapse : the French GINECO - NiQoLe Study
Brief Title: NIraparib and Quality of LifE is a Longitudinal Study Evaluating in Real Life the Tolerability of Niraparib.
Acronym: NiQoLe
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Collaborators: Tesaro, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GINECO-OV239B; 2018-002274-44 (EudraCT Number)
Record Dates: First submitted 2018-11-12; First posted 2018-11-23 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Anti-PARP (poly-ADP ribose polymerase); Late Relapse
MeSH Terms: conditions — Ovarian Neoplasms | interventions — niraparib

STUDY DESIGN:
Masking Description: Open
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NIRAPARIB (Experimental): Oral Niraparib Daily
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — Two different doses of Niraparib can be administrated:
  For patient who had at baseline (T0) a body weight ≥ 77 kg and a platelet count ≥ 150 000/µL, Niraparib will be administrated at a dose of 300 mg daily. The planned dose of 300 mg daily will be made up of three 100 mg capsules.
  For patient who had at baseline (T0) a body weight < 77 kg or a platelet count <150 000/µL, Niraparib will be administrated at a dose of 200 mg daily. The planned dose of 200 mg daily will be made up of two 100 mg capsules.
  Patient should continue to receive study treatment until disease progression as per RECIST as assessed by the investigator or they do not meet any other discontinuation criteria.

SUMMARY:
This is a longitudinal, national, open, multi-centre phase IV study which will recruit up to 141 patients with ovarian cancer in late relapse treated with niraparib according to the labelling In France.

DETAILED DESCRIPTION:
The aim of NiQoLe, phase IV study is to evaluate tolerability of Niraparib and the management by the physicians of the side-effects in real life in France. The study will also generate complementary data of NOVA trial on longitudinal follow up of closed symptoms and side effects reported by the patients especially with the NCI PRO (Patient-Reported Outcome)-CTCAE system. Specific oncogeriatric data will be collected among on a subgroup of elderly patients.

ELIGIBILITY:
Inclusion Criteria:

I-1 Female patients must be ≥ 18 years of age. I-2 Signed informed consent and ability to comply with treatment and follow-up. I-3 Patients with histologically proved high grade epithelial ovarian cancer or fallopian tube or primary peritoneal adenocarcioma.

I-4 Platine sensitive and ovarian, fallopian or peritoneal cancer recurrent patients with a complete response or partial response after a line of platine based chemotherapy.

I-5 Participant must have adequate organ function, defined as follows:

* Absolute neutrophil count ≥ 1,500/μL
* Platelets ≥ 100,000/μL
* Hemoglobin ≥ 9 g/dL
* Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥ 30 mL/min using the Cockcroft-Gault equation
* Total bilirubin ≤ 1.5 x ULN (≤2.0 in patients with known Gilberts syndrome) OR direct bilirubin ≤ 1 x ULN
* Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 x ULN unless liver metastases are present, in which case they must be ≤ 5 x ULN I-6 Patients with an indication of maintenance by Niraparib after platine based chemotherapy according to the labelling (see appendix 17).

I-7 As this study will include patients in France, a subject will be eligible in this study only if either affiliated to, or a beneficiary of, a social category.

I-8 Participant must have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.

I-9 Participant receiving corticosteroids may continue as long as their dose is stable for least 4 weeks prior to initiating protocol therapy.

I-10 Participant must agree to not donate blood during the study or for 90 days after the last dose of Niraparib.

I-11 Female participant has a negative urine or serum pregnancy test within 7 days prior to taking study treatment if of childbearing potential and agrees to abstain from activities that could result in pregnancy from screening through 1 month after the last dose of study treatment, or is of nonchildbearing potential.

I-12 Participant must agree to not breastfeed during the study or for 1 month after the last dose of Niraparib.

I-13 Participant must have normal blood pressure or adequately treated and controlled hypertension

Exclusion Criteria:

E-1 Known hypersensitivity or allergy to active principle or to any components or excipients of the Niraparib formulation.

E-2 Participant must not be simultaneously enrolled in any interventional clinical trial.

E-3 Participant must not have had major surgery ≤ 3 weeks prior to initiating protocol therapy and participant must have recovered from any surgical effects.

E-4 Participant must not have received investigational therapy ≤ 4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is shorter, prior initiating protocol therapy.

E-5 Participant last treatment with platinum-based chemotherapy was ≥12 weeks from initiation of protocol therapy E-6 Participant has had radiation therapy encompassing >20% of the bone marrow within 2 weeks; or any radiation therapy within 1 week prior to Day 1 of protocol therapy.

E-7 Participant must not have received a transfusion (platelets or red blood cells) ≤ 4 weeks NiQoLe - Study protocol - v3.0 on 08/10/2020 Page 10 on 109 N° EudraCT: 2018-002274-44 prior to initiating protocol therapy. E-8 Participant must not have received colony stimulating factors (e.g., granulocyte colonystimulating factor, granulocyte macrophage colony stimulating factor, or recombinant erythropoietin) within 4 weeks prior initiating protocol therapy. E-9 Participant has had any known Grade 3 or 4 anemia, neutropenia or thrombocytopenia due to prior chemotherapy that persisted > 4 weeks and was related to the most recent treatment. E-10 Participant must not have any known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML). E-11 Participant must not have a serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 90 days) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent. E-12 Participant must not be deprived of liberty, under guardianship or under trusteeship.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
Toxicities inducing dose modifications of Niraparib between the start to the cycle 3 (interruption, discontinuation and dose reduction). | 3 months
  Evaluate treatment toxicities

SECONDARY OUTCOMES:
Self-reported fatigue by patient by FACT-F questionnaire (Functional Assessment of Cancer Therapy General - Fatigue) | Up to 18 months.
  Functional Assessment of Cancer Therapy General Fatigue questionnaire (score range from 0 to 52 - Higher scores represent better quality of life)
Self-reported symptoms and side effects with the NCI PRO-CTCAE | Up to 18 months.
  Self-reported symptoms and side effects
Reasons of the dose modification of Niraparib | Up to 18 months.
  Reasons of the dose modification of Niraparib
General health-related quality of life by FACT-G questionnaire (Functional Assessment of Cancer Therapy General) | Up to 18 months.
  Functional Assessment of Cancer Therapy General questionnaire (score range from 0 [worse outcome] to 108 [better outcome])
Pain related to the treatment by Visual Analogic Scale (VAS) | Up to 18 months.
  Score range from 0 [worse outcome] to 10 [better outcome])
Side effects of interest (HTA, anemia, thrombocytopenia) | Up to 18 months.
  Side effects of interest (HTA, anemia, thrombocytopenia)
Duration of Niraparib treatment | Up to 18 months.
  From the start of Niraparib until progression or unacceptable toxicity.
Time to first subsequent line of anti-cancer therapy | Up to 18 months.
  From the stop of Niraparib to the first subsequent line of anti-cancer therapy.
Overall response rate | Up to 18 months.
  Overall response rate
Initial cognitive functions by FACT-cog (Functional Assessment of Cancer Therapy - Cognitive Function) questionnaire | At the inclusion visit
  FACT-cog questionnaire (score range from 0 to 132 - Higher scores represent better functioning)
Plasma level of Niraparib before Niraparib administration | Day 8
  residual dosage of Niraparib
Plasma level of Niraparib before Niraparib administration | 3 months
  residual dosage of Niraparib
Geriatric Depression Scale (score range from 0 [better outcome] to 30 [worse outcome]) | Up to 6 months.
  Geriatric Depression Scale (score range from 0 [better outcome] to 30 [worse outcome])

CONTACTS AND LOCATIONS:
Overall Officials: Florence JOLY, MD, PhD, Principal Investigator — Centre François Baclesse 3, avenue du Général Harris 14076 CAEN
Locations (30):
- France (30):
  - Sainte-Catherine Institut du Cancer Avignon-Provence, Avignon
  - Centre Hospitalier de la Côte Basque, Bayonne
  - CHRU Jean Minjoz, Besançon
  - Clinique Tivoli, Bordeaux
  - Institut Bergonié, Bordeaux
  - Hôpital Fleyriat, Bourg-en-Bresse
  - Centre François Baclesse, Caen
  - Medipole de Savoie, Challes-les-Eaux
  - SASU Centre d'Oncologie et Radiothérapie 37, Chambray-lès-Tours
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges François Leclerc, Dijon
  - Groupe Hospitalier Mutualiste de Grenoble - Institut Daniel Hollard, Grenoble
  - Les Hôpitaux de Chartres - Hôpital Louis Pasteur, Le Coudray
  - Hôpital Privé Jean Mermoz, Lyon
  - ICM Val d'Aurelle, Montpellier
  - Médipôle de NANCY / Centre d'Oncologie de Gentilly, Nancy
  - Centre Antoine Lacassagne, Nice
  - Centre ONCOGARD - Institut de Cancérologie du Gard, Nîmes
  - Centre Hospitalier Régional d'Orléans, Orléans
  - Hôpital Cochin, Paris
  - Groupe Hospitalier Diaconesses-Croix Saint Simon, Paris
  - Centre CARIO - HPCA, Plérin
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Institut du Cancer Courlancy, Reims
  - Clinique Mutualiste de l'Estuaire, Saint-Nazaire
  - CHU de Saint-Etienne - Pôle de Cancérologie, Saint-Priest-en-Jarez
  - Centre Hospitalier Saint-Malo, St-Malo
  - Hôpitaux Universitaires de Strasbourg - Institut de Cancérologie Strasbourg Europe, Strasbourg
  - Clinique Pasteur, Toulouse
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy

REFERENCES:
- [Derived] Joly F, Bazan F, Garbay D, Ouldbey Y, Follana P, Champeaux-Orange E, Legouffe E, Brachet PE, Spaeth D, Combe P, Hardy-Bessard AC, Selle F, Grenier J, Lebreton C, Derbel O, Bonnet E, Fournel P, Fernandez Diez Y, Delecroix V, Emambux S, Alexandre J, Grellety T, Mille D, Orfeuvre H, Favier C, Le Roux D, Mouret-Reynier MA, Quesada S, Kurtz JE. Improving real-world evaluation of patient- and physician-reported tolerability: niraparib for recurrent ovarian cancer (NiQoLe). JNCI Cancer Spectr. 2025 Jan 3;9(1):pkae114. doi: 10.1093/jncics/pkae114. PMID 39673810